CLINICAL TRIAL: NCT01516658
Title: Efficacy of Hydrogel Coil on Endovascular Treatment for Intracranial Aneurysms; Multi-center, Prospective, Randomized, Open-label Blind-endpoint Trial
Brief Title: HYdrogel Coil Versus Bare Platinum Coil in Recanalization Imaging Data Study
Acronym: HYBRID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kobe City General Hospital (Other)
Collaborators: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Principal Investigator, Nobuyuki Sakai, Director of Neurosurgery, Kobe City General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIBRAIN1119; UMIN000006748 (Other: UMIN Japan)
Record Dates: First submitted 2011-11-29; First posted 2012-01-25 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Intracranial Aneurysm; Subarachnoid Hemorrhage
Keywords: intracranial aneurysm; endovascular therapy; detachable coil; recanalization
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrogel coil group (Experimental): use Hydrogel Coil as much as be able to use
  Interventions: Device: Hydrogel coil
- Bare platinum coil group (Active Comparator): use only bare platinum coil
  Interventions: Device: Bare platinum coil

INTERVENTIONS:
Device: Hydrogel coil — at least one Hydrogel coil have to use for embolization
  Other Names: Hydrocoil; HydroSoft; HydroFrame
  Arms: Hydrogel coil group
Device: Bare platinum coil — only bare platinum coil have to use for embolization
  Other Names: detachable coil; GDC; Microvention
  Arms: Bare platinum coil group

SUMMARY:
HYBRID study is prospective randomized open label controlled multi center trial, to compare Hydrocoil and bare platinum coil for recanalization after endovascular treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
At least one Hydrocoil have to use in Hydrocoil arm, and only bare platinum coil have to use in Control arm.

Primary endpoint is recanalization within 1 year after embolization, and secondary endpoint are:

1. aneurysmal rupture within 1 year after embolization
2. any event within 30 days after embolization
3. recanalization within 6 months after embolization
4. aneurysmal retreatment within 1 year after embolization
5. aneurysmal rupture and any death within 1 year after embolization
6. any stroke within 1 year after embolization
7. any stroke, death hemorrhagic event, aneurysmal recanalization or retreatment within 1 year after embolization
8. change in aneurysmal occlusion
9. any comlicaion within 1 year after embolization
10. %length of Hydrocoil, maximum diameter of aneurysm, volume embolization ratio.

ELIGIBILITY:
Inclusion Criteria:

* saccular intracranial aneurysm
* endovascular treatment scheduled within 60days after consent
* 20-79 years old
* unruptured, chronic SAH or acurte SAH Grade 1-III
* 7-20mm in size
* 1 year follow up possibel
* independent (mRS 0-2)
* document consent

Exclusion Criteria:

* previous endovascular treated
* additional aneurysm scheduled of endovascular treatment
* pregnant
* ineligible for study

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
recanalization within 1 year after embolization | 1 year

SECONDARY OUTCOMES:
aneurysmal rupture within 1 year after embolization | 1 year
any event within 30 days after embolization | 30 days
aneurysmal retreatment within 1 year after embolization | 1 year
aneurysmal rupture and any death within 1 year after embolization | 1 year
any stroke within 1 year after embolization | 1 year
any stroke, death hemorrhagic event, aneurysmal recanalization or retreatment within 1 year after embolization | 1 year
change in aneurysmal occlusion | 1 year
any complicaion within 1 year after embolization | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sakai, MD, DMSc, Principal Investigator — Kobe City Medical Center General Hospital
Locations (2):
- Japan (2):
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - Kobe City General Hospital, Kobe, Hyōgo